CLINICAL TRIAL: NCT06973018
Title: Internetförmedlad Kognitiv Rehabilitering Vid Lindrig Kognitiv störning
Brief Title: Internet Delivered Cognitive Rehabilitation for Mild Cognitive Impairments
Acronym: eRehabCog
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Aniko Bartfai (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Sponsor-Investigator, Aniko Bartfai, senior professor in neuropsychology, Karolinska Institutet, Danderyd Hospital
Organization: Danderyd Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dnr 202003079
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Traumatic Brain Injury; Stroke; Multiple Sclerosis; Parkinsons Disease (PD); Post-COVID-19 Condition
Keywords: brain injury; cognitive rehabilitation; nervous system disorders; eHealth; self assessment
MeSH Terms: conditions — Brain Injuries, Traumatic; Stroke; Multiple Sclerosis; Parkinson Disease; Brain Injuries; Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: Participating teams were randomized to either of the two intervention arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eRehabCog (Experimental): 10 week (1 hour / week, 10 hours in total) internet delivered manualised cognitive rehabilitation
  Interventions: Behavioral: eRehabCog
- CogMed QM (Active Comparator): 5 week (2 hours / week, 10 hours in total) internet delivered working memory training program
  Interventions: Behavioral: CogMed QM

INTERVENTIONS:
Behavioral: eRehabCog — eRehabCog is a manualised internet delivered compensatory cognitive rehabilitation program (10 weeks, 1 hour per week, 10 hours in total). It is designed to improve patient self efficacy and participation in everyday life activities through compensatory strategy learning
  Arms: eRehabCog
Behavioral: CogMed QM — CogMed QM is an internet delivered training program (5 weeks, 2 hours per week, 10 hours in total) designed to improve patients working memory
  Arms: CogMed QM

SUMMARY:
Acquired brain injury and neurological disorders cause cognitive deficits, which in turn cause reduced participation in everyday life. Cognitive rehabilitation, where patients learn about cognition, cognitive deficits and ways to circumvent problems arising from deficits can increase participation and quality of life. ERehabCog is an internet delivered cognitive rehabilitation program intended for patients suffering mild to moderate impairments. The program consists of information and homework assignments, which take approximately 10 weeks to complete with the assistance of a therapist. Effects are evaluated through measures of everyday life participation, mood, and life satisfaction and compared with an attention training program. This study aims to contribute to the evidence base for internet delivered cognitive rehabilitation for mild to moderate cognitive impairments. Evidence based interventions are vital to use the potential of technology to the benefit of affected patients.

DETAILED DESCRIPTION:
When broadly defined, diseases and injuries affecting the central nervous system are one of the leading causes of disease burden in the world affecting more than 3 billion people. With such a large proportion of the global population affected, optimization of limited resources in the form of specialized rehabilitation is instrumental to ensuring sustainable public health.

The consequences of acquired brain injuries (ABIs) and neurological disorders are multifaceted, causing diminished functional capacity in a range of areas. Cognitive impairments are common, affecting ability to work, take on reponsibilities at home and in the community. Relationships in all significant life areas can be disrupted. As a result, patients may experience a significant shift in a plurality of life roles. Rehabilitation aims to help patients recapture premorbid capacities and reduce the impact of deficits while considering the needs and context of the patient. Cognitive rehabilitation has the potential to ameliorate patient outcomes. Patients in Sweden are offered cognitive rehabilitation as a part of multimodal rehabilitation programs, typically provided in university hospital settings. The demand for such interventions is greater than the amount provided. Patients with mild cognitive deficits are generally less prioritized than those with greater impairments. Internet provided rehabilitation programs can increase the accessibility of cognitive rehabilitation.

eRehabCog is an internet-delivered 10 module cognitive rehabilitation program designed to aid patients experiencing mild to moderate cognitive deficits following acquired brain injury or neurological disorders. The philosophy behind the development of eRehabCog is grounded in a compensatory-metacognitive approach. That is to say, patients learn about cognitive functions, consequences of deficits and ways to compensate. This approach has both a practical component where patients learn strategies they may use in their everyday life and a self-reflective component where patients learn to think about their thinking in such a way to raise their awareness of their functioning.

CogMed QM is a 10 week digital working memory training program which has been evaluated in children with ADHD and adults with stroke, showing improvements in working memory function. CogMed QM is a restitutive training program, intended to help patients retake diminished working memory capacity.

The overall aim of this study is to evaluate the efficacy of eRehabCog for patients experiencing mild to moderate cognitive deficits. Specific aims are to 1) evaluate the efficacy of eRehabCog for patients with ABI and ND admitted to community neurorehabilitation 2) compare the effects of eRehabCog to CogMed QM

The study will recruit 64 patients enrolled in community neurorehabilitation. Patients recruited will be ≥ 18 years old, have obtained a score ≥ 21 on Montreal Cognitive Assessment (MoCA), living in their home, with our without assistance and with access to computer and/or functionally ecquivalent device. Exclusion criteria will be progressive neurocognitive impairment (i.e dementia), substance abuse, insufficient Swedish language capabilities, insufficiently stable living situation to commit to a 10 week long program. Community neurorehabilitation teams participating in the study will be randomized to either eRehabCog or CogMed QM.

The primary outcome measure is the Mayo Portland Adaptability Inventory - Fourth edition (MPAI-4) Participation.

Secondary outcome measures are MPAI-4 Total score, ability and adjustment, Hospital Anxiety and Depression Scale (HADS), Life Satisfaction Scale - 11 items (LiSat-11), Community Integration Questionnaire - revised (CIQ-R) and Patient Satisfaction Questionnaire (PSQ).

Background information on patients general status including socioeconomic factors and medical factors such as time since diagnosis is also collected. Behavioural measures such as time in the program, amount of messages to therapist and number of logins are additionally collected throughout participation.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in community neurorehabilitation in Stockholm, Sweden
* Mild to moderate cognitive impairment as a consequence of acquired brain injury or nervous system disease
* MoCA 21 ≥
* Sufficient command of Swedish language
* Access to internet connected device and internet connection

Exclusion Criteria:

* Severe and enduring psychiatric or behavioural disorders (i.e Schizophrenia, substance abuse)
* Suspected or diagnosed dementia
* Homelessness or other social instability rendering access to internet unpredictable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2021-05-02 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Mayo Portland Adaptability Inventory - fourth edition (MPAI-4), Participation subscale | Two weeks before intervention, at intervention start, at the end of treatment at 10 weeks, at six months post intervention ed
  Change in T-score

SECONDARY OUTCOMES:
MPAI-4 Adaptability subscale | Two weeks before intervention, at intervention start, at the end of treatment at 10 weeks, at six months post intervention ed
  Change in T-score
MPAI-4 Abilities subscale | Two weeks before intervention, at intervention start, at the end of treatment at 10 weeks, at six months post intervention ed
  Change in T-score
MPAI-4 Total score | Two weeks before intervention, at intervention start, at the end of treatment at 10 weeks, at six months post intervention ed
  Change in T-score
Hospital Anxiety and Depression Scale | Two weeks before intervention, at intervention start, at the end of treatment at 10 weeks, at six months post intervention ed
  Change in average total score
Life Satisfaction Questionnaire (LiSat-11) | Two weeks before intervention, at intervention start, at the end of treatment at 10 weeks, at six months post intervention ed
  Change in average total score
Community Integration Questionnaire - Revised (CIQ-R) | Two weeks before intervention, at intervention start, at the end of treatment at 10 weeks, at six months post intervention ed
  Change in total and subscale scores

OTHER OUTCOMES:
Patient satisfaction questionnaire | End of treatment at 10 weeks
  Correlation to primary and secondary outcome measures
Montreal Cognitive Assessment (MoCA) | Baseline
  Correlation to primary and secondary outcome measures

CONTACTS AND LOCATIONS:
Overall Officials: Aniko Bartfai, PhD, Principal Investigator — Karolinska Institutet Danderyds Sjukhus (KIDS), Department of medical rehabilitation
Locations (1):
- Danderyd Hospital, Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No
According to the decision of the ethical review board, IPD can not be shared.

REFERENCES:
- See also: Description of eRehabCog in text and video format (Swedish) — https://www.ds.se/ditt-besok/undersokning-och-behandling/rehabilitering/erehabcog/
- See also: Description of Cogmed QM from company webpage (English and Swedish) — https://www.cogmed.com/